CLINICAL TRIAL: NCT00995358
Title: Phase II Multicenter Trial of Peptide Vaccination Therapy Using Novel Cancer Testis Antigens for Locally Advanced, Recurrent, or Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: A Study With Peptide Vaccination in Treating Patients With Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Yamanashi (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: First Department of Surgery, University of Yamanashi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMU-02
Record Dates: First submitted 2009-10-08; First posted 2009-10-15 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Esophageal Cancer
Keywords: Epitope peptide; CTL; Esophageal cancer; Vaccination
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Peptides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vaccination (Experimental)
  Interventions: Biological: peptide

INTERVENTIONS:
Biological: peptide — Each of three peptides (1mg) mixed with IFA (1ml) were injected every week at five round.

SUMMARY:
The purpose of this study is to evaluate overall survival and immunological monitoring for peptide vaccination therapy using novel cancer testis antigens for locally advanced, recurrent, or metastatic esophageal squamous cell carcinoma (ESCC).

DETAILED DESCRIPTION:
The phase I vaccination study using peptides derived from TTK, LY6K, and IMP-3 for locally advanced, recurrent or metastatic esophageal squamous cell carcinoma (ESCC) who had failed for the standard therapy indicated that the vaccine treatment were well tolerated and feasible, and that antigen-specific T cell responses were strongly induced by the vaccination with some objective clinical responses. Thus, we are currently initiating the randomized phase II clinical vaccination study for the same cohort with ESCC to evaluate the survival benefit of the cancer vaccination.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS

* Locally advanced, recurrent or metastatic esophageal squamous cell carcinoma who had failed for the standard therapy

PATIENTS CHARACTERISTICS

* ECOG performance status 0-2
* Age≧ 20≦ 80years
* WBC≥ 2,000/mm³ Platelet count ≥ 75,000/mm³ Total bilirubin ≤ 2.0 x the institutional normal upper limits AST, ALT, ALP ≤ 2.5 x the institutional normal upper limits Creatinine ≤ 1.5 x the institutional normal upper limits
* No therapy 4 weeks prior to the initiation of the trial
* Able and willing to give valid written informed consent

Exclusion Criteria:

* Pregnancy (women of childbearing potential: Refusal or inability to use effective means of contraception)
* Breastfeeding
* Serious bleeding disorder
* Serious infections requiring antibiotics
* Concomitant treatment with steroids or immunosuppressing agent
* Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival after the 1st vaccination | 2 years

SECONDARY OUTCOMES:
Antigen specific control response induced by vaccination | 1 year
DTH response induced by vaccination | 1 year
Time to progression after the 1st vaccination | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Koji Kono, MD.PhD, Principal Investigator — University of Yamanashi, First Deparment of Surgery
Locations (1):
- First Department of Surgery, University of Yamanashi, Chūō, Yamanashi, Japan

REFERENCES:
- [Result] 1. Okabe H, Satoh S, Kato T, et al. Genome-wide analysis of gene expression in human hepatocellular carcinomas using cDNA microarray: identification of genes involved in viral carcinogenesis and tumor progression. Cancer Res 2001; 61: 2129-37. 2 Lin YM, Furukawa Y, Tsunoda T, Yue CT, Yang KC, Nakamura Y. Molecular diagnosis of colorectal tumors by expression profiles of 50 genes expressed differentially in adenomas and carcinomas. Oncogene 2002; 21: 4120-28. 3. Hasegawa S, Furukawa Y, Li M, et al. Genome-wide analysis of gene expression in intestinal-type gastric cancers using a complementary DNA microarray representing 23,040 genes. Cancer Res 2002; 62: 7012-17. 4. Suda T, Tsunoda T, Daigo Y, Nakamura Y, Tahara H. Identification of human leukocyte antigen-A24-restricted epitope peptides derived from gene products upregulated in lung and esophageal cancers as novel targets for immunotherapy. Cancer Sci 2007; 98: 1803-8. 5. Ishikawa N, Takano A, Yasui W, et al. Cancer-testis antigen lymphocyte antigen 6 complex locus K is a serologic biomarker and a therapeutic target for lung and esophageal carcinomas. Cancer Res 2007; 67: 11601-11. 6. Yoshiki Mizukami, Koji Kono, Yataro Daigo, et al. Detection of novel Cancer-Testis antigen-specific T-cell responses in TIL, regional lymph nodes and PBL in patients with esophageal squamous cell carcinoma. Cancer Science 2008 ;99:1448-54 6. Koji Kono, Yoshiki Mizukami, Yataro Daigo, Atsushi Takano, Ken Masuda, Koji Yoshida, Takuya Tsunoda, Yoshihiko Kawaguchi, Yusuke Nakamura, and Hideki Fujii. Vaccination with Multiple Peptides derived from Novel Cancer-Testis Antigens Can Induce Specific T-Cell Responses and Clinical Responses in Advanced Esophageal cancer. Cancer Sci. 2009;100:1502-9.
- [Derived] Kono K, Iinuma H, Akutsu Y, Tanaka H, Hayashi N, Uchikado Y, Noguchi T, Fujii H, Okinaka K, Fukushima R, Matsubara H, Ohira M, Baba H, Natsugoe S, Kitano S, Takeda K, Yoshida K, Tsunoda T, Nakamura Y. Multicenter, phase II clinical trial of cancer vaccination for advanced esophageal cancer with three peptides derived from novel cancer-testis antigens. J Transl Med. 2012 Jul 9;10:141. doi: 10.1186/1479-5876-10-141. PMID 22776426